CLINICAL TRIAL: NCT00100178
Title: New Onset of Type 1 Diabetes Mycophenolate Mofetil-Daclizumab Clinical Trial (Preservation of Pancreatic Production of Insulin Through Immunosuppression-POPPII #1)
Brief Title: New Onset of Type 1 Diabetes Mycophenolate Mofetil-Daclizumab Clinical Trial
Acronym: TN02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Juvenile Diabetes Research Foundation (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TN02 MMF/DZB; U01DK061055 (NIH); UC4DK097835 (NIH)
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: immunosuppressive therapy; Type 1 Diabetes TrialNet; TrialNet; POPPII; POPPII-1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Daclizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MMF and DBZ (Experimental): DZB given by intravenous infusion (1 mg/kg)at baseline and 2 weeks later, and MMF given orally at dose of 600 mg/m2 (2000 mg/day maximum) in 2-3 divided doses for 2 years.
  Interventions: Drug: Mycophenolate mofeteil (MMF); Drug: Daclizumab (DZB)
- MMF Alone (Experimental): MMF given orally at dose of 600 mg/m2 (2000 mg/day maximum) in 2-3 divided doses for 2 years and saline intravenous infusions given at baseline and two weeks later.
  Interventions: Drug: Mycophenolate mofeteil (MMF); Drug: Placebo control for Daclizumab (DZB)
- Placebo (Placebo Comparator): Placebo pills given daily for two years and saline intravenous infusions given at baseline and two weeks later.
  Interventions: Drug: Placebo control for Mycophenolate mofeteil (MMF); Drug: Placebo control for Daclizumab (DZB)

INTERVENTIONS:
Drug: Mycophenolate mofeteil (MMF)
  Arms: MMF Alone; MMF and DBZ
Drug: Daclizumab (DZB)
  Arms: MMF and DBZ
Drug: Placebo control for Mycophenolate mofeteil (MMF) — Placebo pills taken orally
  Arms: Placebo
Drug: Placebo control for Daclizumab (DZB) — saline intravenous infusions
  Arms: MMF Alone; Placebo

SUMMARY:
The objective of this study is to identify immune intervention strategies that will preserve residual beta cell function at the onset of type 1 diabetes. Scientific evidence developed over the last 10 - 20 years suggests that type 1 diabetes is a chronic, slowly progressive autoimmune disease and that clinical symptoms do not develop until at least 80% - 90% of beta cell mass has been destroyed as a result of the autoimmune process. It is now recognized that preservation of remaining beta cells is clinically important as the ability to secrete, even small amounts of insulin, can make the disease easier to control and help minimize complications associated with having years of inadequate glycemic control.

This clinical trial is the first in a series of studies to be launched by the TrialNet Study Group to test various interventions for preserving residual beta cell function in new onset type 1 diabetes. Specifically, this study is designed to determine the ability of Mycophenolate Mofetil (MMF/CellCept) used alone, or in combination with Daclizumab (DZB/Zenapax) to see if it is possible to stop the immune system from destroying beta cells in new onset type 1 diabetes patients (within 3 months of diagnosis.)

Researchers have made great strides in understanding how the immune system works and in changing the activity of immune cells with medicines called immunotherapies. Some immunotherapies work by making the immune system less active. Scientists have discovered that key immune cells, called T cells, help to cause type 1 diabetes. These T cells are largely responsible for attacking the beta cells that produce insulin. Doctors have found medicines that slow or suppress the activity of T cells. It is hoped that these immunosuppressive medicines can help treat type 1 diabetes by stopping T cells before they destroy all of the beta cells.

Medicines that make the immune system less active have been developed and studied for other diseases. Mycophenolate mofetil (MMF) and Daclizumab (DZB) are two of these medicines. Their effects on the immune system are well understood. Researchers believe these medicines may lessen the immune system's destruction of beta cells that leads to type 1 diabetes. In addition, researchers hope the effect of these medicines will last longer than other therapies.

The goal of this study is to find out if two medicines are able to stop the ongoing destruction of beta cells which are still functioning at the time type 1 diabetes is diagnosed. The two immunosuppressive medications being tested are Mycophenolate mofetil (MMF/CellCept®) and Daclizumab (DZB/Zenapax®). They work by making the immune system less active. TrialNet researchers hope that these medications will help maintain insulin secretion from remaining beta cells and thus help to maintain better glycemic control. Even if the medications work, study participants will still need to take insulin injections but it may make it easier to control normal blood sugar levels which can help reduce long-term complications of diabetes such as blindness, kidney failure, nerve damage, heart attack and stroke.

The aim is to arrest beta cell destruction in newly diabetic subjects because immune modulation may not work well alone once the autoimmune process has progressed to complete or near complete destruction of beta cells. The study's rationale is to demonstrate a meaningful preservation of islet function with minimal immune system side effects over the 4-year course of this study.

The data from this clinical trial could serve as the basis for a larger trial if the results are sufficiently positive, or they could suggest other combined intervention trials that might achieve either better efficacy or potentially preserve C-peptide without the need for continued immunosuppression.

DETAILED DESCRIPTION:
Design of Study:

The study is a multi-center, three-arm, randomized, double-masked, placebo-controlled clinical trial. Comparisons will be made among the three groups, which are:

* Mycophenolate mofetil active drug with Daclizumab (DZB) placebo IV
* Mycophenolate mofetil active drug with active Daclizumab IV
* Mycophenolate mofetil placebo with Daclizumab placebo IV

Participants that agree to enroll in the study will be asked to take study medications for two years. MMF is given by mouth twice a day. DZB is given by an intravenous infusion twice, once at the time of enrollment and again two weeks later. Both these medications are approved by the U.S. Food and Drug Administration and are used by people who have received an organ transplant. This study is testing a new use of these medications to preserve insulin secretion by delaying or stopping further destruction of insulin-secreting cells in people with newly diagnosed type 1 diabetes. Both MMF and DZB make the immune system less active. Participants will be monitored closely for any possible side effects that can occur from taking either DZB and/or MMF due to decreased activity of the immune system.

Participants will need to go to the Clinical Center for visits and tests. For the first month participants will come in every week; then participants will come in at month 2 and month 3. After the month 3 visit, visits will occur about every three months. At most visits, blood will be drawn and participants will meet with a study physician to review their overall diabetes management, and be monitored for any possible side-effects from the study medication.

Participants will be asked to do a longer test called a Mixed Meal Tolerance Test (MMTT) at the initial visit and at five additional visits while taking the assigned study medication. The MMTT involves drinking a special drink which has a controlled amount of carbohydrates, protein, and fat to measure residual insulin secretion. The test requires having an IV inserted into the arm and having blood samples taken from the IV over a period of 2 to 4 hours. After completing the two year period of taking the study medication, participants will be asked to return every 3-6 months for an additional 1-2 years to evaluate their ability to secrete insulin after discontinuing the study medication.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must meet the following inclusion criteria:

* Be within 3-months of diagnosis of type 1 diabetes based on American Diabetes Association (ADA) criteria
* Be between the ages of 8 and 45 years old
* Must have stimulated C-peptide levels > 0.2 pmol/ml (measured during an MMTT administered no more than one month prior to the date of randomization)
* Must have either detectable anti-GAD, anti-ICA512/IA-2, insulin autoantibodies (unless received insulin therapy for 7 days or more), or islet cell autoantibodies.

[The reason for inclusion of these enrollment criteria is to avoid inclusion of patients with "Type 1B diabetes mellitus", which may not involve the immunologic criteria measured by the assays that will be utilized.]

* If participant has reproductive potential, he or she must be agreeable to an effective form of birth control (unless abstinence is the chosen method).
* If participant is female with reproductive potential, she must be willing to undergo pregnancy testing and to report possible or confirmed pregnancies promptly during the course of the MMF/DZB study.
* Must be willing to comply with intensive diabetes management. The goal of management will be an HbA1c of 7.0% for all participants, regardless of age. Participants will be expected to take a sufficient number of daily insulin shots to meet this goal. Alternatively, participants can use insulin pump therapy. Participants will also be expected to test their blood sugar at least 3-4 times per day. There will be a Certified Diabetes Educator working with study participants to achieve these goals.

Exclusion Criteria:

Potential participants must not meet any of the following exclusion criteria:

* Have any complicating medical issues that would interfere with blood drawing or monitoring.
* Have a Body Mass Index (BMI) that is greater than the 95th percentile for age and gender.
* Have serologic evidence of HIV infection.
* Have serologic evidence of Hepatitis B infection.
* Have serologic evidence of Hepatitis C infection.
* Have abnormal liver function tests.
* Have a history of leukopenia and/or neutropenia.
* Have a history of chronic peptic ulcer disease, erosive esophagitis, chronic inflammatory bowel disease and/or chronic colonic disease.
* Have a positive PPD test result.
* Have had any live vaccinations in the preceding 6 weeks (e.g. MMR-second dose, live flu vaccine, varicella vaccine, live polio vaccine, yellow fever vaccine).
* Resides outside reasonable geographical proximity to the clinic (i.e., residence outside the state in which the Investigator and study reside, residence outside an immediately neighboring state, or residence outside an area that the Investigator considers reasonable). It is left to the Investigator's discretion to decide if a patient's geographical residence is prohibitive to complete study participation.
* Require chronic use of steroids or other immunosuppressive agents for other conditions.
* Be currently pregnant or 3 months postpartum.
* Be currently nursing or within 6 weeks of having completed nursing.
* Anticipate getting pregnant, or fathering a child, during the study.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2004-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Skyler, M.D., Study Chair — University of Miami
Locations (11):
- United States (10):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California-San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Benaroya Research Institute, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/tn02-mmfdzb/?query=tn02
URL: https://repository.niddk.nih.gov/studies/tn02-mmfdzb/?query=tn02

REFERENCES:
- [Background] Palmer JP, Fleming GA, Greenbaum CJ, Herold KC, Jansa LD, Kolb H, Lachin JM, Polonsky KS, Pozzilli P, Skyler JS, Steffes MW. C-peptide is the appropriate outcome measure for type 1 diabetes clinical trials to preserve beta-cell function: report of an ADA workshop, 21-22 October 2001. Diabetes. 2004 Jan;53(1):250-64. doi: 10.2337/diabetes.53.1.250. PMID 14693724
- [Background] Kaufman DB, Leventhal JR, Stuart J, Abecassis MM, Fryer JP, Stuart FP. Mycophenolate mofetil and tacrolimus as primary maintenance immunosuppression in simultaneous pancreas-kidney transplantation: initial experience in 50 consecutive cases. Transplantation. 1999 Feb 27;67(4):586-93. doi: 10.1097/00007890-199902270-00017. PMID 10071032
- [Background] Feutren G, Papoz L, Assan R, Vialettes B, Karsenty G, Vexiau P, Du Rostu H, Rodier M, Sirmai J, Lallemand A, et al. Cyclosporin increases the rate and length of remissions in insulin-dependent diabetes of recent onset. Results of a multicentre double-blind trial. Lancet. 1986 Jul 19;2(8499):119-24. doi: 10.1016/s0140-6736(86)91943-4. PMID 2873396
- [Background] Placebo-controlled study of mycophenolate mofetil combined with cyclosporin and corticosteroids for prevention of acute rejection. European Mycophenolate Mofetil Cooperative Study Group. Lancet. 1995 May 27;345(8961):1321-5. PMID 7752752
- [Background] Brazelton TR, Morris RE. Molecular mechanisms of action of new xenobiotic immunosuppressive drugs: tacrolimus (FK506), sirolimus (rapamycin), mycophenolate mofetil and leflunomide. Curr Opin Immunol. 1996 Oct;8(5):710-20. doi: 10.1016/s0952-7915(96)80090-2. PMID 8902398
- [Result] Gottlieb PA, Quinlan S, Krause-Steinrauf H, Greenbaum CJ, Wilson DM, Rodriguez H, Schatz DA, Moran AM, Lachin JM, Skyler JS; Type 1 Diabetes TrialNet MMF/DZB Study Group. Failure to preserve beta-cell function with mycophenolate mofetil and daclizumab combined therapy in patients with new- onset type 1 diabetes. Diabetes Care. 2010 Apr;33(4):826-32. doi: 10.2337/dc09-1349. Epub 2010 Jan 12. PMID 20067954
- [Derived] Loechelt BJ, Boulware D, Green M, Baden LR, Gottlieb P, Krause-Steinrauf H, Weinberg A; Type 1 Diabetes TrialNet Daclizumab/Mycophenolic Acid Study Group. Epstein-Barr and other herpesvirus infections in patients with early onset type 1 diabetes treated with daclizumab and mycophenolate mofetil. Clin Infect Dis. 2013 Jan;56(2):248-54. doi: 10.1093/cid/cis848. Epub 2012 Oct 5. PMID 23042974
- See also: TrialNet Study Group — http://www.diabetestrialnet.org
- See also: American Diabetes Association — http://www.diabetes.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen Clinical Centers at academic institutions recruited and enrolled 126 subjects ages 8 to 45 years with autoimmune T1D for less than 3 months.
Pre-assignment Details: Subjects were screened for evidence of autoantibodies and c-peptide >0.2 pmol on a stimulated 2 hr Mixed Meal Tolerance Test to determine eligibility for the study.The MMTT must be conducted at least 21 days from the diagnosis of diabetes and no more than one month (37 days) prior to the date of randomization.
Groups:
- MMF and DZB: DZB given by intravenous infusion (1 mg/kg)at baseline and 2 weeks later, and 600 mg/m2 (2000 mg/day maximum) in 2-3 divided doses for 2 years.
- MMF Alone: 600 mg/m2 (2000 mg/day maximum) in 2-3 divided doses for 2 years and saline intravenous infusions given at baseline and two weeks later.
- MMF-DZB Placebo Control: Placebo pills given daily for two years and saline intravenous infusions given at baseline and two weeks later.
Period: Overall Study
Arm/Group | MMF and DZB | MMF Alone | MMF-DZB Placebo Control
Started | 41 | 31 (12 subjects randomized to the MMF alone group were excluded from analysis due to randomization error) | 42
Completed | 32 | 21 | 32
Not Completed | 9 | 10 | 10
Not completed — Lost to Follow-up | 0 | 6 | 5
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Physician Decision | 6 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- MMF and DZB: 600 mg/m2 (2000 mg/day maximum) in 2-3 divided doses for 2 years AND DZB given by intravenous infusion (1 mg/kg)at baseline and 2 weeks later.
- Total: Total of all reporting groups
Arm/Group | MMF and DZB | MMF Alone | MMF-DZB Placebo Control | Total
Number analyzed (Participants) | 41 | 31 | 42 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.4 (9.09) | 17.1 (6.71) | 18.8 (10.44) | 18.2 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 17 | 46
  Male | 23 | 20 | 25 | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Stimulated C-peptide Area Under the Curve
Description: The primary outcome is the area under the stimulated C-peptide curve (AUC) based on data collected at time 0 to 2 hours of a 4-hour mixed meal glucose tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30 60, 90, and 120 minutes.
Time Frame: 2 years
Population: Participants who completed a 4-hour mixed meal glucose tolerance test at the two-year visit were included in the analysis
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ml
Groups:
- Placebo Control: Placebo pills given daily for two years and saline intravenous infusions given at baseline and two weeks later.
Arm/Group | MMF and DZB | Placebo Control | MMF Alone
Number analyzed (Participants) | 22 | 20 | 18
pmol/ml | 0.28 [0.19 to 0.37] | 0.27 [0.18 to 0.37] | 0.25 [0.14 to 0.37]
Statistical Analysis 1: Comparison: MMF and DZB vs Placebo Control; The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis; Test type: Superiority or Other; p = 0.47, ANCOVA

ADVERSE EVENTS:
Groups:
- MMF and DZB: 600 mg/m2 (2000 mg/day maximum) in 2-3 divided doses for 2 years and DZB given by intravenous infusion (1 mg/kg)at baseline and 2 weeks later .
Arm/Group | MMF and DZB | MMF Alone | MMF-DZB Placebo Control
Serious Adverse Events (participants affected / at risk) | 15/41 | 5/31 | 5/42
Other Adverse Events (participants affected / at risk) | 41/41 | 31/31 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMF and DZB (N=41) | MMF Alone (N=31) | MMF-DZB Placebo Control (N=42)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood/Bone Marrow Unspecified (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Laboratory Unspecified (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mood alteration (Psychiatric disorders) | 1 (2) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary Malignancy Unspecified (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal- Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMF and DZB (N=41) | MMF Alone (N=31) | MMF-DZB Placebo Control (N=42)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 2 (3) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 6 (7) | 0 (0) | 3 (3)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 4 (5) | 5 (10) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5 (7) | 4 (10) | 0 (0)
Blood/Bone Marrow Unspecified (Blood and lymphatic system disorders) | 6 (9) | 7 (14) | 7 (13)
Vasovagal episode (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (4) | 3 (4) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (7) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 (14) | 3 (5) | 5 (6)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4) | 0 (0)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Dental: periodontal disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dental: teeth (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (14) | 5 (8) | 12 (13)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (6)
Nausea (Gastrointestinal disorders) | 7 (11) | 5 (5) | 6 (7)
Vomiting (Gastrointestinal disorders) | 8 (11) | 7 (8) | 6 (6)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 0 (0) | 3 (5) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 5 (6) | 4 (4) | 5 (6)
Infection - Other (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 10 (18) | 6 (15) | 7 (8)
Infection with unknown ANC (Infections and infestations) | 36 (106) | 27 (61) | 34 (94)
Infection Unspecified (Infections and infestations) | 10 (23) | 2 (11) | 6 (8)
Lymphatics - Other (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 13 (24) | 9 (21) | 10 (26)
Metabolic/Laboratory Unspecified (Metabolism and nutrition disorders) | 8 (10) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 7 (8)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 8 (13) | 3 (5) | 9 (10)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Mood alteration (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Other AE Unspecified (General disorders) | 5 (6) | 5 (11) | 5 (8)
Pain (General disorders) | 10 (11) | 6 (18) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 2 (2) | 4 (5)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 0 (0)
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3)
Flu-like syndrome (General disorders) | 0 (0) | 0 (0) | 4 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No